CLINICAL TRIAL: NCT03939000
Title: Clinical Profile and Laboratory Finding of Diabetic Foot Ulcers From Tertiary Hospitals in Bali
Brief Title: Clinical Profile and Laboratory Finding of DFU From Tertiary Hospitals in Bali
Status: Completed | Type: Observational
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Hendry Irawan, General Surgeon, Udayana University
Other Study IDs: Profile_DFU
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Foot Ulcer; Type 2 Diabetes Mellitus; Laboratory Problem; Physical Findings.Skin Ulcer
Keywords: clinical profile; diabetic foot ulcer; laboratory finding; tertiary hospital
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2; Skin Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators want to obtain the clinical profile, hematological profile, and biochemical profile from diabetic foot ulcer (DFU) patient.

DETAILED DESCRIPTION:
This study is a retrospective descriptive study reviewing the medical records of diabetic foot patients who were admitted to Sanglah General Hospital for surgical procedure. Sanglah General Hospital is a provincial hospital located in Denpasar, Bali, which is the central referral hospital in Bali and Nusa Tenggara islands as known as a tertiary hospital.

All DFU patients who underwent surgical procedures in Sanglah General Hospital operating theatre were included in the study. All patient medical records were provided by our hospital information center system. A diagnosis of diabetes mellitus was defined and confirmed from ICD (International Classification of Diseases)-10 code E11.622 for "Type 2 Diabetes Mellitus with other skin ulcers".

Data which we collected from the hospital information center system were further addressed into different aspects, which comprised of personal data, DFU severity, diabetes mellitus duration, ulcer duration, treatment procedures, and laboratory results. Based on our main objective of this study, we divide the laboratory results into two groups, hematological and blood chemistry profile. The variables selected in the hematological profile were hemoglobin, hematocrit, leukocyte and differential counts, and platelet. The variables which were included in blood chemistry profile are alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum albumin, random blood glucose, glycated hemoglobin (HbA1c), blood urea nitrogen (BUN), serum creatinine, serum sodium, serum potassium, prothrombin time (PTT), activated partial thromboplastin time (APTT), and international normalized ratio (INR).

The protocol of DFU management in our hospital included diagnosis and treatment of infection (local and systemic), assessment of patient's diabetic status, treatment of infection, diabetes mellitus, and wound care, and also surgical procedure, such as sharp debridement and amputations. The procedures were classified into five categories, consist of debridement, amputation of the fingers, transmetatarsal amputation, amputation below the knee, and amputation above the knee. DFU severity is classified into five different grades, based on Wagner's diabetic foot classification. In our hospital, patients with diabetic foot problems were evaluated and treated by a team consisting of surgeons, endocrinologists, microbiologists, rehabilitation specialists, nutritionists, and nurses.

For the statistical analyses, variables were assessed using the program IBM SPSS statistics version 23.0 for Windows (IBM Corporation, New York, USA). All numerical data were summarized as mean ± standard deviation, and categorical variables were summarized as frequency and percentage. Our method is about to use every available data to descriptively picture laboratory characteristics in DFU patients.

ELIGIBILITY:
Inclusion Criteria:

* DFU patients who underwent surgical procedures in Sanglah General Hospital operating theatre.

Exclusion Criteria:

* DFU patients without surgical intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All DFU patients who underwent surgical procedures in Sanglah General Hospital operating theatre.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Age | Before surgery
  Age in years
Diabetes mellitus duration | Before surgery
  Diabetes mellitus duration in years
Foot ulcer duration | Before surgery
  Foot ulcer duration in weeks
Gender | Before surgery
  Gender is classified to male and female
Foot affected | Before surgery
  Foot affected is classified to right foot, left foot, and bilateral
Wagner classification | Before surgery
  Wagner classification is classified to grade 1, grade 2, grade 3, grade 4, and grade 5
Surgical procedure | After surgery
  Surgical procedure is classified to debridement, finger amputation, transmetatarsal amputation, below the knee amputation, and above the knee amputation
Hemoglobin | Before surgery
  Hemoglobin in g/dL
Hematocrit | Before surgery
  Hematocrit in %
Leukocyte | Before surgery
  Leukocyte in 10^9/L
Basophil | Before surgery
  Basophil in 10^9/L
Eosinophil | Before surgery
  Eosinophil in 10^9/L
Neutrophil | Before surgery
  Neutrophil in 10^9/L
Lymphocyte | Before surgery
  Lymphocyte in 10^9/L
Monocyte | Before surgery
  Monocyte in 10^9/L
Platelet | Before surgery
  Platelet in 10^9/L
Alanine aminotransferase | Before surgery
  Alanine aminotransferase (ALT) in U/L
Aspartate aminotransferase | Before surgery
  Aspartate aminotransferase (AST) in U/L
Serum albumin | Before surgery
  Serum albumin in g/dL
Random blood glucose | Before surgery
  Random blood glucose in mg/dL
Glycated hemoglobin | Before surgery
  Glycated hemoglobin (HbA1c) in %
Blood urea nitrogen | Before surgery
  Blood urea nitrogen (BUN) in mg/dL
Serum creatinine | Before surgery
  Serum creatinine in mg/dL
Serum sodium | Before surgery
  Serum sodium in mmol/L
Serum potassium | Before surgery
  Serum potassium in mmol/L
Prothrombin time | Before surgery
  Prothrombin time (PT) in seconds
Activated partial thromboplastin time | Before surgery
  Activated partial thromboplastin time (APTT) in seconds
International normalized ratio | Before surgery
  International normalized ratio (INR) has no units (it is a ratio) and is determined to decimal place. INR formula is (patient PT/mean normal PT)ISI.
  ISI stands for International Sensitivity Index

REFERENCES:
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Zimmet PZ, Alberti KG. Epidemiology of Diabetes-Status of a Pandemic and Issues Around Metabolic Surgery. Diabetes Care. 2016 Jun;39(6):878-83. doi: 10.2337/dc16-0273. PMID 27222545
- [Background] Balducci S, Sacchetti M, Haxhi J, Orlando G, D'Errico V, Fallucca S, Menini S, Pugliese G. Physical exercise as therapy for type 2 diabetes mellitus. Diabetes Metab Res Rev. 2014 Mar;30 Suppl 1:13-23. doi: 10.1002/dmrr.2514. PMID 24353273
- [Background] Kayssi A, Rogers LC, Neville RF. General Considerations in Diabetic Foot Ulcers. In: Sidawy AN and Perler BA, editors. Rutherford's Vascular Surgery and Endovascular Therapy. 9th ed. Philadelphia: Elsevier Inc; 2019. p.1514-26.
- [Background] International Diabetes Federation. IDF Clinical Practice Recommendations on the Diabetic Foot - 2017: A guide for healthcare professionals. Brussels: International Diabetes Federation; 2017.
- [Background] Pemayun TGD, Naibaho RM. Diabetes Management Diabetic Foot Ulcer Registry at a Tertiary Care Hospital in Semarang, Indonesia: an Overview of its Clinical Profile and Management Outcome. J Clin Diabetes Pract. 2016;1:111.
- [Background] Leong M, Murphy KD, Phillips LG. Wound Healing. In: Townsend Jr CM, Beauchamp RD, Evers BM, Mattox KL, editors. Sabiston Textbook of Surgery: The Biological Basis of Modern Surgical Practice. 20th ed. Philadelphia: Elsevier Inc; 2017. p.130-62.
- [Background] Barbul A, Efron DT, Kavalukas SL. Wound Healing. In: Brunicardi FC, Andersen DK, Billiar TR, et al, editors. Schwartz Principles of Surgery. 10th ed. New York: McGraw Hill Education; 2015. p. 241-71.
- [Background] Kratz A, Ferraro M, Sluss PM, Lewandrowski KB. Case records of the Massachusetts General Hospital. Weekly clinicopathological exercises. Laboratory reference values. N Engl J Med. 2004 Oct 7;351(15):1548-63. doi: 10.1056/NEJMcpc049016. No abstract available. PMID 15470219
- [Background] Powers AC. Diabetes Mellitus. In: Longo DL, Fauci AS, Kasper DL, Hauser SL, Jameson JL, Loscalzo J, editors. Harrison's Principles of Internal Medicine. 18th ed. New York: McGraw Hill Education; 2011. p.2968-2970.
- [Background] Viswanathan V, Thomas N, Tandon N, Asirvatham A, Rajasekar S, Ramachandran A, Senthilvasan K, Murugan VS, Muthulakshmi. Profile of diabetic foot complications and its associated complications--a multicentric study from India. J Assoc Physicians India. 2005 Nov;53:933-6. PMID 16515230
- [Background] Tarigan TJE, Yunir E, Subekti I, Pramono LA, Martina D. Profile and analysis of diabetes chronic complications in Outpatient Diabetes Clinic of Cipto Mangunkusumo Hospital, Jakarta. Med J Indones. 2015;24:156-62.
- [Background] Pemayun TG, Naibaho RM, Novitasari D, Amin N, Minuljo TT. Risk factors for lower extremity amputation in patients with diabetic foot ulcers: a hospital-based case-control study. Diabet Foot Ankle. 2015 Dec 7;6:29629. doi: 10.3402/dfa.v6.29629. eCollection 2015. PMID 26651032
- [Background] Bowker JH. Minor and Major Lower-Limb Amputations and Disarticulations in Patients with Diabetes Mellitus. In: Bowker JH, Pfeifer MA. Levin and O'Neal's the Diabetic Foot. 7th ed. Philadelphia: Elsevier Inc; 2008. p.403-28.
- [Background] Demirdal T, Sen P. The significance of neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and lymphocyte-monocyte ratio in predicting peripheral arterial disease, peripheral neuropathy, osteomyelitis and amputation in diabetic foot infection. Diabetes Res Clin Pract. 2018 Oct;144:118-125. doi: 10.1016/j.diabres.2018.08.009. Epub 2018 Sep 1. PMID 30176260
- [Background] Metineren H, Dulgeroglu TC. Comparison of the Neutrophil/Lymphocyte Ratio and C-Reactive Protein Levels in Patients With Amputation for Diabetic Foot Ulcers. Int J Low Extrem Wounds. 2017 Mar;16(1):23-28. doi: 10.1177/1534734617696729. Epub 2017 Mar 8. PMID 28682678
- [Background] Balta S, Celik T, Mikhailidis DP, Ozturk C, Demirkol S, Aparci M, Iyisoy A. The Relation Between Atherosclerosis and the Neutrophil-Lymphocyte Ratio. Clin Appl Thromb Hemost. 2016 Jul;22(5):405-11. doi: 10.1177/1076029615569568. Epub 2015 Feb 9. PMID 25667237
- [Background] Goldman MP, Clark CJ, Craven TE, Davis RP, Williams TK, Velazquez-Ramirez G, Hurie JB, Edwards MS. Effect of Intensive Glycemic Control on Risk of Lower Extremity Amputation. J Am Coll Surg. 2018 Dec;227(6):596-604. doi: 10.1016/j.jamcollsurg.2018.09.021. Epub 2018 Oct 16. PMID 30336205
- [Background] Bhonsle HS, Korwar AM, Kote SS, Golegaonkar SB, Chougale AD, Shaik ML, Dhande NL, Giri AP, Shelgikar KM, Boppana R, Kulkarni MJ. Low plasma albumin levels are associated with increased plasma protein glycation and HbA1c in diabetes. J Proteome Res. 2012 Feb 3;11(2):1391-6. doi: 10.1021/pr201030m. Epub 2012 Jan 6. PMID 22181049
- [Background] Shatnawi NJ, Al-Zoubi NA, Hawamdeh HM, Khader YS, Garaibeh K, Heis HA. Predictors of major lower limb amputation in type 2 diabetic patients referred for hospital care with diabetic foot syndrome. Diabetes Metab Syndr Obes. 2018 Jun 22;11:313-319. doi: 10.2147/DMSO.S165967. eCollection 2018. PMID 29950877
- [Background] Kahraman C, Yümün G, Kahraman NK, Namdar ND, Cosgun S. Neutrophil-to-lymphocyte ratio in diabetes mellitus patients with and without diabetic foot ulcer. Eur J Med Sci. 2014;1:8-13.
- [Background] Vatankhah N, Jahangiri Y, Landry GJ, McLafferty RB, Alkayed NJ, Moneta GL, Azarbal AF. Predictive value of neutrophil-to-lymphocyte ratio in diabetic wound healing. J Vasc Surg. 2017 Feb;65(2):478-483. doi: 10.1016/j.jvs.2016.08.108. Epub 2016 Nov 23. PMID 27887858
- [Background] Semadi IN, Irawan H. Blood glucose and lipid profile in patients with diabetic foot ulcer that underwent hyperbaric oxygen therapy. Bali Med J. 2017;6:405-8.
- [Background] Irawan H, Semadi IN, Widiana IGR. A Pilot Study of Short-Duration Hyperbaric Oxygen Therapy to Improve HbA1c, Leukocyte, and Serum Creatinine in Patients with Diabetic Foot Ulcer Wagner 3-4. ScientificWorldJournal. 2018 Aug 12;2018:6425857. doi: 10.1155/2018/6425857. eCollection 2018. PMID 30158840
- [Background] Wounds International. International Best Practice Guidelines: Wound Management in Diabetic Foot Ulcers. London: Wounds International A division of Schofield Healthcare Media Limited Enterprise House; 2013.
- [Background] Waniczek D, Kozowicz A, Muc-Wierzgon M, Kokot T, Swietochowska E, Nowakowska-Zajdel E. Adjunct methods of the standard diabetic foot ulceration therapy. Evid Based Complement Alternat Med. 2013;2013:243568. doi: 10.1155/2013/243568. Epub 2013 Jun 13. PMID 23843866